CLINICAL TRIAL: NCT04073654
Title: Clinical Evaluation and Primary Stability of Early Loaded Implants With Sandblasted and Acid-etched Surface Versus Implants With SA Surface Modified With pH Buffering Agent: a Multicenter Randomized Controlled Trial
Brief Title: SA Versus SOI Surfaces for Single Implant-supported Crown
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osstem AIC (Other)
Responsible Party: Principal Investigator, Marco Tallarico, Coordinator, Osstem AIC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOI_1_RCT_MT
Record Dates: First submitted 2019-06-27; First posted 2019-08-29 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Dental Implant Failed; Bone Resorption
Keywords: Dental implants; Implant surfaces; Marginal bone loss
MeSH Terms: conditions — Bone Resorption | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, split-mouth design
Who Masked: Participant, Outcomes Assessor
Masking Description: Implants have same macro design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SA Implants (Active Comparator): Dental implant with sandblasted and Acid-etched (SA) surface
  Interventions: Procedure: Placement of dental implants (surgical procedure)
- SOI Implants (Experimental): Same dental implant with sandblasted and Acid-etched surface modified with pH buffering agent
  Interventions: Procedure: Placement of dental implants (surgical procedure)

INTERVENTIONS:
Procedure: Placement of dental implants (surgical procedure) — The two study implants have to be placed in the same surgical session according to similar procedures. Implants will be placed in the planned anatomic sites by using a flapless or a miniflap approach. Implants sites will be prepared based on the bone density, and according to the manufacturers's instruction by using the 122 Taper kit (Osstem Implant).

SUMMARY:
The purpose of this randomized controlled trial is to compare clinical data and implant stability of immediately loaded TSIII Osstem implants with Sandblasted and Acid-etched (SA) surface versus implants with SA surface modified with pH buffering agent for the rehabilitation of single implant-supported crown.

DETAILED DESCRIPTION:
This study aimed to evaluate if there are some benefits using novel implant surface. This surface should improve the secondary implant stability, reducing the overall time needed for the osseointegration. main benefits in clinical practice should be reduced treatment time.

ELIGIBILITY:
Inclusion Criteria:

* Any partially edentulous subject requiring at least two single (preferable non-adjacent) implant-supported crowns, being at least 18 year old and able to sign an informed consent will be screened for eligibility. Bone volumes should allow the placement of two implants at least 8.5 mm (maximum 10 mm) long and 4.5 mm (minimum 3.5 mm) wide, with a minimal insertion torque of 30 Ncm. Implants can be placed in previous post-extractive socket or in augmented bone, if at least 4 to 6 months have passed from the extraction or from augmentation procedures.

Exclusion Criteria:

* Patients unable to commit to 5 years follow-up.
* General contraindications to implant surgery.
* Less then 4 mm of keratinised gingiva crestally (at the implant sites).
* Immune-suppressed/compromised patients.
* Patients irradiated in the head and/or neck.
* Uncontrolled diabetes.
* Pregnancy or lactation.
* Untreated periodontal disease.
* Poor oral hygiene and motivation (full mouth bleeding and full mouth plaque index higher than 25%).
* Addiction to alcohol or drugs.
* Psychiatric problems and/or unrealistic expectations.
* Patients with an acute infection or suppuration in the site intended for implant placement.
* Patients needing any form of tissue augmentation at implant placement.
* Immediate post-extractive implants (implants can be placed after a 3-month healing period).
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* Patients referred only for implant placement if the follow-up cannot be done at the treatment center.
* Patients participating in other studies, if the present protocol could not be fully adhered to.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Implant failure | From implant placement up to 60 months after loading
  Implant removal for any reason will be considered an implant failure.
Crown failure | From crown delivery up to 60 months
  Crown replacement for any reason will be considered a crown failure.
Complications | From implant placement up to 60 months after loading
  Any complications will be recorded. Examples of biological complications are: nerve injury, fistula, peri-implantitis. Examples of biomechanical complications are fracture of the abutments screw, loosening of the crown, fracture of the ceramic.

SECONDARY OUTCOMES:
Peri-implant marginal bone level (MBL) changes | From implant placement up to 60 months after loading
  It will be assessed on periapical radiographs taken with the paralleling technique. The distance between marginal bone level and implant/abutment junction, will be measured at both mesial and distal sides and averaged. Bone level changes at single implants will be averaged at group level. Non-digital radiographs will be scanned, digitized, and stored in a personal computer. Peri-implant marginal bone levels will be measured using the Scion Image (Scion Corporation, Frederick, MD, USA) software. The software will be calibrated for every single image using the known distance of the implant neck. Measurements of the mesial and distal bone crest level adjacent to each implant will be made to the nearest 0.01 mm. Reference points for the linear measurements will be: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact.
Probing pocket depth (PPD) | From crown delivery up to 60 months
  Probing pocket depth will be measured by a blinded operator, with a periodontal probe (PCP-UNC 15, Hu-Friedy Manufacturing, Chicago, IL, USA). Three vestibular and three lingual values will be collected and averaged for each implant.
Bleeding on probing (BOP) | From crown delivery up to 60 months
  Bleeding on probing will be measured by a blinded operator, with a periodontal probe (PCP-UNC 15, Hu-Friedy Manufacturing, Chicago, IL, USA). Three vestibular and three lingual values will be collected and averaged for each implant.
plaque index (PI) | From implant placement up to 60 months after loading
  Plaque index will be measured by a blinded operator, with a periodontal probe (PCP-UNC 15, Hu-Friedy Manufacturing, Chicago, IL, USA) at delivery of the definitive crowns, 1, 3, and 5 years follow-up in function. Three vestibular and three lingual values will be collected for each implant.
Implant stability quotient | The ISQ values will be recorded at the time of implant placement (baseline) and then 1,2,3,4,5,6,7,8, and 12 weeks after implant placement.
  The implant stability quotient will be recorded by the blind outcome assessor using resonance frequency analysis (Osstell Mentor; Osstell, Goteborg, Sweden).7 Buccopalatal and mesiodistal measurements will be taken and averaged, with the result being displayed by the device in ISQ units, ranging from 1 to 100.
Pink Esthetic Score | From crown delivery up to 60 months
  The aesthetic evaluation will be performed according to the pink aesthetic score on the vestibular and occlusal pictures taken including at least one adjacent tooth per side.8 The values will be assessed at definitive prosthesis delivery, and then early up to the end of the follow-up. Seven variables (mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture) will be assessed with a 2-1-0 score (2 being best and 0 being poorest) by the same blinded dentist.

CONTACTS AND LOCATIONS:
Locations (10):
- Erta Xhanari, Tirana, Albania
- Elitsa Deliverska, Sofia, Bulgaria
- Italy (3):
  - Fulvio Gatti, Milan
  - Studio Odontoiatrico Marco Tallarico, Rome
  - Leonardo Muzzi, Siena
- Łukasz Zadrożny, Warsaw, Poland
- Cesaltino Remedios, Fátima, Portugal
- Mircea, Craiova, Romania
- Andre de Waal, South Africa, South Africa
- Nicolas Widmer, Bern, Switzerland